CLINICAL TRIAL: NCT02450656
Title: Phase I/II Study With the Combination of Afatinib and Selumetinib in Advanced KRAS Mutant Positive and PIK3CA Wildtype Non-small Cell Lung Cancer
Brief Title: Afatinib and Selumetinib in Advanced KRAS Mutant and PIK3CA Wildtype Non-small Cell Lung Cancer
Acronym: M14AFS
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: AstraZeneca (Industry); Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: M14AFS
Record Dates: First submitted 2014-11-13; First posted 2015-05-21 (Estimated); Last update posted 2018-08-27 (Actual); Status verified 2018-08

CONDITIONS: Colorectal Neoplasms; Gastrointestinal Neoplasms; Pancreatic Neoplasms; Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Colorectal Neoplasms; Gastrointestinal Neoplasms; Pancreatic Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Afatinib; AZD 6244; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Afatinib plus selumetinib (Experimental): Combination of afatinib and selumetinib at the optimal dose and regimen as determined in the phase I part of this study
  Interventions: Drug: Afatinib; Drug: Selumetinib
- Control (Active Comparator): Standard-of-care second line treatment for non small cell lung cancer (docetaxel)
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Afatinib — Tablet
  Other Names: BIBW2992
  Arms: Afatinib plus selumetinib
Drug: Selumetinib — Capsule
  Other Names: AZD6244
  Arms: Afatinib plus selumetinib
Drug: Docetaxel
  Arms: Control

SUMMARY:
This is a multi-center open-label proof-of-concept study consisting of two parts: PART A - a phase I dose-finding study (3 + 3 classical design) evaluating the RP2D of afatinib in combination with selumetinib in KRASm NSCLC; and PART B - a randomized phase II study investigating the progression free survival and safety of selumetinib/afatinib combination therapy compared to standard of care chemotherapy in KRASm NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological proof of advanced NSCLC; for PART B: treated with first line therapy for metastatic disease only.
* Written documentation of a known pathogenic KRAS (exon 2, 3 or 4) mutation and PIK3CA wildtype (defined as absence of mutations in exon 9 and 20)
* Able and willing to give written informed consent
* Able and willing to undergo blood sampling for PK and PD analysis
* Life expectancy >=3 months allowing adequate follow up of toxicity evaluation and antitumor activity.
* WHO performance status of 0 or 1.
* Able and willing to undergo a tumor biopsies prior to start, after two weeks (part A only) and upon progression of disease
* Measurable disease according to RECIST 1.1
* Adequate organ system function measured by laboratory values

Exclusion Criteria:

* Any treatment with investigational drugs within 30 days prior to receiving the first dose of investigational treatment.
* History of another malignancy Exception PART A: Patients who have been disease-free for at least 3 years, or patients with a history of completely resected non-melanoma skin cancer and/or patients with indolent second malignancies are eligible. Exception PART B: Adequately treated carcinoma in situ of the cervix and adequately treated basal cell carcinoma of the skin. 3. Symptomatic or untreated leptomeningeal disease.
* Symptomatic brain metastasis.
* Patients previously treated with any drug combination known to interfere with EGFR, HER2, HER3, HER4 or MAPK- and PI3K-pathway components, including inhibitors of PTEN, PI3K, AKT, mTOR, BRAF, MEK and ERK.
* History of interstitial lung disease or pneumonitis
* Radio-, immuno- or chemotherapy within the last 2 weeks prior to receiving the first dose of investigational treatment. Palliative radiation (1x 8Gy) is allowed.
* Opthalmological diseases
* Patients with left ventricular ejection fraction (LVEF) < 55%
* Patients with cardiac comorbidities
* Concomitant or recent use (in the past 14 days) of strong inhibitors and inducers of CYP1A2, CYP2C19, CYP3A4, 3A5 and P-glycoprotein (P-gp)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2015-06; Primary Completion 2019-05 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicities (Phase I) | Cycle 1 (4 weeks)
  Incidence of DLTs in the first treatment cycle
Progression Free Survival (Phase II) | CT scan every 6 weeks and monthly phone call until start of subsequent anticancer therapy or until all patients have been followed up for at least 18 months of have been lost to follow up, whichever occurs first
  PFS measured by RECIST v 1.1

SECONDARY OUTCOMES:
Tolerability (Incidence and severity of adverse events per CTCAE v4.03) | Up to 28 days after last study drug intake
  Incidence and severity of adverse events per CTCAE v4.03
Plasma concentrations of afatanib and selumetinib | On day 1, 2, 4, 8, 15, 22 in cycle 1, on day 1 and 2 in cycle 2 and subsequently at every treatment cycle pre-dose
  Plasma concentrations of afatanib and selumetinib will be measured at day 1,2,4,8,15, 22 in cycle 1, on day 1 and 2 in cycle 2 and subsequently before every treatment cycle to determine pharmacokinetics of both substances in combination and interindividual differences after a single dose and after multiple doses.
Efficacy (Phase II) (Overall response rate (ORR), duration of response (DOR) , time to response (TTR) and overall survival (OS) per RECIST v1.1) | Assessed by CT scans every 6 weeks and by monthly phone call until all patients have been followed up for at least 18 months or have been lost to follow up, whichever occurs first.
  Overall response rate (ORR), duration of response (DOR) , time to response (TTR) and overall survival (OS) per RECIST v1.1

OTHER OUTCOMES:
Determinants and mode of response - Target proteins | At baseline, cycle 1 day 15 and at treatment discontinuation (expected 6-9 months after start)
  Change in expression and/or phosphorylation status target proteins (e.g. pERK, pS6, heregulin, HER2) before, during and after treatment
Pharmacogenetics profiling to assess predictors of response and resistance- inducing mutations | Before treatment, every 6 weeks and at treatment discontinuation (expected 6-9 months after start)
  Pharmacogenetic profiling to assess predictors of response and resistance- inducing mutations

CONTACTS AND LOCATIONS:
Overall Officials: F Opdam, MD, PhD, Principal Investigator — NKI-AvL
Locations (2):
- Netherlands (2):
  - UMC St. Radboud Nijmegen, Nijmegen, Gelderland
  - Netherlands Cancer Institute - Antoni van Leeuwenhoek Hospital, Amsterdam